CLINICAL TRIAL: NCT00001094
Title: A Phase II, Randomized, Controlled, Open-Label Trial of Combination Therapy With Nelfinavir (NFV) and Saquinavir (SQV)Sgc With Delavirdine (DLV) or 3TC/ZDV Versus Nelfinavir (NFV) and 3TC/ZDV in Subjects With HIV Infection and > 5,000 HIV RNA Copies/ML
Brief Title: A Comparison of Nelfinavir Plus Saquinavir Plus Delavirdine or 3TC/ZDV Versus Nelfinavir Plus 3TC/ZDV in HIV-Infected Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 374
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; Zidovudine; Lamivudine; RNA, Viral; Saquinavir; Delavirdine; Anti-HIV Agents; Nelfinavir
MeSH Terms: conditions — HIV Infections | interventions — lamivudine, zidovudine drug combination; Nelfinavir; Saquinavir; Delavirdine

INTERVENTIONS:
Drug: Lamivudine/Zidovudine
Drug: Nelfinavir mesylate
Drug: Saquinavir
Drug: Delavirdine mesylate

SUMMARY:
To compare the long-term virologic response to combination therapy with two protease inhibitors, i.e., nelfinavir (NFV) + saquinavir soft gel capsule (SQVsgc) and delavirdine (DLV) or combination lamivudine/zidovudine (3TC/ZDV, Combivir) versus NFV and 3TC/ZDV, in the proportion of patients demonstrating virologic success (< 500 copies/ml HIV RNA) at week 48, without prior virologic or clinical failure. To evaluate the safety and tolerance of combination protease inhibitors.

To evaluate the durability of virologic response as assessed by the Roche Ultra Sensitive assay (< 200 copies/ml) and culturable virus. To compare time to a confirmed virologic response (two consecutive plasma HIV RNA levels < 500 copies/ml) or to a confirmed treatment relapse following a confirmed virologic response across the treatment arms. To evaluate biologic phenotype (non-syncytium inducing versus syncytium inducing capacity) and the evolution and patterns of viral resistance among patients with confirmed treatment failures at or after weeks 16 to 24. To compare immunologic benefits, as measured by longitudinal CD4/CD8 cell count profiles. To evaluate the influence of baseline virologic and immunologic parameters on the magnitude and duration of plasma HIV RNA response. To compare virologic response between the two dose schedules of NFV and SQVsgc (bid vs tid) and between NFV and SQVsgc with either DLV or combination 3TC/ZDV. To evaluate compliance and exploratory population pharmacometrics.

Past studies have shown that combination therapies not only will result in better clinical outcomes but may prolong the effects of therapy. The enhanced effects seen with combination therapies are likely related to a greater suppression of HIV replication and alterations in resistance patterns. Both in vitro and in vivo studies suggest that triple-drug therapy may have an advantage over one- and two-drug regimens. Therefore, triple-drug therapy appears to be an important strategy in the treatment of HIV infection.

DETAILED DESCRIPTION:
Past studies have shown that combination therapies not only will result in better clinical outcomes but may prolong the effects of therapy. The enhanced effects seen with combination therapies are likely related to a greater suppression of HIV replication and alterations in resistance patterns. Both in vitro and in vivo studies suggest that triple-drug therapy may have an advantage over one- and two-drug regimens. Therefore, triple-drug therapy appears to be an important strategy in the treatment of HIV infection.

This is a Phase II, randomized, controlled, open-label trial of NFV + SQVsgc and either DLV or combined 3TC/ZDV versus NFV and combined 3TC/ZDV. Prior to randomization, patients are stratified by HIV RNA (above or below 65,000 copies/ml) and by prior antiretroviral therapy (no therapy vs any therapy). Patients (100 patients/arm) are then randomly assigned to one of four arms. Arm I receives NFV plus combination 3TC/ZDV. Arm II receives NFV plus SQVsgc plus combination 3TC/ZDV. Arm III receives NFV plus SQVsgc plus DLV. Arm IV receives NFV plus SQVsgc plus DLV. Treatment continues for 48 weeks following enrollment of the last patient. Response to treatment is assessed at week 16. Patients with confirmed plasma HIV RNA levels >= 500 copies/ml at week 16 whose plasma HIV RNA has decreased since study entry (day 0) may continue therapy and be reassessed at weeks 20 and 24. Patients considered treatment failures (i.e., 2 consecutive plasma HIV RNA levels >= 500 copies/ml at or after week 16) or who have relapsed may register to Step 2 treatment (addition of at least 2 new drugs to their prior treatment regimen), enroll in another ACTG protocol at time of failure, or seek the best available therapy while continuing to be followed for remainder of study.

ELIGIBILITY:
This study has been terminated.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fischl M, Study Chair; Bartlett J, Study Chair
Locations (17):
- United States (16):
  - Willow Clinic, Menlo Park, California
  - Stanford Univ Med Ctr, Stanford, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Univ of Miami School of Medicine, Miami, Florida
  - Emory Univ, Atlanta, Georgia
  - Queens Med Ctr, Honolulu, Hawaii
  - Univ of Hawaii, Honolulu, Hawaii
  - Louis A Weiss Memorial Hosp, Chicago, Illinois
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Carolinas Med Ctr, Charlotte, North Carolina
  - Moses H Cone Memorial Hosp, Greensboro, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Univ of Texas Galveston, Galveston, Texas
- Univ of Puerto Rico, San Juan, Puerto Rico